CLINICAL TRIAL: NCT02892435
Title: Wound Healing After Dirty/Contaminated Emergency Abdominal Surgery: Prevena™ Incision Management System vs Conventional Management
Brief Title: Prevena™ Incision Management System vs Conventional Management for Wound Healing
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Marco Scatizzi, Chief, general surgery department, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 012/2015
Record Dates: First submitted 2015-05-19; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Wound Healing; Prevena; Dirty Abdominal Surgery; Contaminated Abdominal Surgery; Emergency Abdominal Surgery; Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena arm (Experimental): patients underwent to contaminated/dirty surgery who positioned incisional negative pressure wound therapy and kept for six days
  Interventions: Device: incisional negative pressure wound therapy
- Control arm (Active Comparator): patients underwent to contaminated/dirty surgery who positioned conventional dressing
  Interventions: Device: conventional dressing

INTERVENTIONS:
Device: incisional negative pressure wound therapy — positioning incisional negative pressure therapy over closed wound.
  Other Names: Prevena - KCI
  Arms: Prevena arm
Device: conventional dressing — positioning conventional dressing
  Arms: Control arm

SUMMARY:
Comparison in abdominal wound healing after contaminated or dirty surgery with incisional negative pressure wound therapy versus standard dressing.

DETAILED DESCRIPTION:
All patients submitted to contaminated or dirty abdominal surgery have more risk of surgical site infections. The investigators intend to randomize this kind of patients and comparison wound healing after dressed with incisional negative pressure wound therapy or standard dressing.

In the study group INPWT (Prevena) is positioned immediately next surgery and dressed for six days. Every patients will be medicate in sixth, ninth, fifteenth and thirtieth day after surgery and will be valued wound healing with a scale score.

Moreover for each patient it will be assessed risk developing wound complications through possum score and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* abdominal surgery
* open surgery
* contaminated or dirty surgery

Exclusion Criteria:

* not abdominal surgery
* mininvasive surgery
* clean surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) reduction | 7 months
  quantify SSI decrease after incisional negative pressure wound therapy

SECONDARY OUTCOMES:
Surgical Site Infection (SSI) and risk factors as diabetis, obesity and cancer | 2 years
  check connection between wound complications and risk factors and showing if Incisional Negative Pressure Wound Therapy (INPWT) could reduce effects of these risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Feroci, MD, Principal Investigator — Ospedale Santo Stefano Prato
Locations (1):
- Misericordia e Dolce Hospital, Prato, Po, Italy

IPD SHARING:
Plan to Share IPD: No